CLINICAL TRIAL: NCT03396458
Title: Prevalence and Risk Factors of Hepatitis B Viral Infection in the Turkish Population Living in Belgium
Brief Title: Hepatitis B Prevalence in the Turkish Population Living in Middle Limburg
Acronym: HBVTR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Clinical Associate Professor, Hasselt University
Other Study IDs: HBVTR-1.0
Record Dates: First submitted 2017-12-15; First posted 2018-01-11 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Disease prevalence; Screening; Migrant; Turkish; Belgium
MeSH Terms: conditions — Hepatitis B | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatitis B group: Hepatitis B serology and questionnaire
  Interventions: Diagnostic Test: Hepatitis B serology; Other: Questionnaire

INTERVENTIONS:
Diagnostic Test: Hepatitis B serology — A serum specimen will be taken and assessed for hepatitis B serology (HBsAg, anti-HBs and anti-HBc).
Other: Questionnaire — Participants will be asked to fill in a questionnaire regarding sociodemographic factors, migration history, risk factors for HBV infection (e.g. sharing toothbrushes, HBV infected family member) and HBV vaccination status.

SUMMARY:
This study will assess HBV (HBsAg, anti-HBc and anti-HBs) prevalence in the Turkish population living in Belgium. Additionally, the investigators will determine the risk factors for HBV infection and the uptake of screening, vaccination and antiviral treatment in this hard-to-reach Turkish population.

DETAILED DESCRIPTION:
HBV infection is an important public health problem in the Turkish population, i.e. one of the largest migrant populations in Europe. With the introduction of cost-effective antiviral treatments in the past decade, there is a need to identify HBV infected patients who may benefit from treatment. This study will assess the HBV prevalence in the Turkish population living in Belgium. Additionally, the investigators will determine the risk factors of HBV infection and the uptake of screening, vaccination and antiviral treatment in this hard-to-reach Turkish population.

A cross-sectional, epidemiological trial will be conducted in the region Middle Limburg Belgium, where the Turkish adult population (subjects born in Turkey or subjects of which one of the parents is born in Turkey), 18 years of age and older, will be screened for HBsAg, anti-HBs and anti-HBc. Educational meetings concerning viral hepatitis B will be organized and there will be three ways to be screened for HBV: (1) immediately after the educational meetings, (2) at the Outpatient Hepatology Department of Ziekenhuis Oost-Limburg (ZOL) and (3) at home visits. Subsequently, participants will be asked to fill in a questionnaire regarding sociodemographic factors, migration history, risk factors for HBV infection (e.g. sharing toothbrushes, HBV infected family member) and HBV vaccination status. One year after data collection, HBsAg positive patients will be assessed whether they are under follow-up at the general practitioner or hepatologist. The investigators will also gather information regarding the uptake of vaccination in non-immunized subjects.

This study will provide information about the HBV prevalence and distribution of the stages of liver disease in the Turkish population in Belgium. By determining the risk factors for HBV infection, subgroups with an increased prevalence of HBV infection can be identified. This study will also give information on how to organize the healthcare system for screening in hard-to-reach migrant groups and to develop care paths.

ELIGIBILITY:
Inclusion Criteria:

* Turkish origin, defined as one of the parents born in Turkey
* Having a signed informed consent form

Exclusion Criteria:

/

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Turkish population
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of current HBV infection in the Turkish population | 1 day
  Serum HBsAg

SECONDARY OUTCOMES:
Seroprevalence of protective antibodies against HBV infection in the Turkish population | 1 day
  Serum anti-HBs
Assess risk factors for past or current HBV infecion in the Turkish population | 1 day
  Combine results from (1) serum anti-HBc with (2) questionnaire regarding sociodemographic factors, migration, risk factors for HBV infection and HBV vaccination status

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, M.D., Ph.D., Principal Investigator — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koc OM, Hens N, Bielen R, Van Damme P, Robaeys G. Hepatitis B virus prevalence and risk factors in hard-to-reach Turkish population living in Belgium: A protocol for screening. Medicine (Baltimore). 2019 May;98(18):e15412. doi: 10.1097/MD.0000000000015412. PMID 31045797